CLINICAL TRIAL: NCT05311553
Title: Zona Pellucida Thinning Versus Drilling During Laser-assisted Hatching of Human Embryos in Intracytoplasmic Sperm Injection
Brief Title: Zona Pellucida Thinning Versus Drilling During Laser-assisted Hatching
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19-121 thinning vs drilling
Record Dates: First submitted 2022-03-27; First posted 2022-04-05 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zona pellucida thinning (Experimental): thinning will be performed without reaching the inner membrane of the Zona pellucida thickness.
  Interventions: Procedure: Zona pellucida thinning
- Zona pellucida drilling (Experimental): an opening will be made from the outside to the inside of the Zona pellucida.
  Interventions: Procedure: Zona pellucida drilling

INTERVENTIONS:
Procedure: Zona pellucida thinning — Laser-assisted hatching will be conducted using a Laser System with a 1.48-μm diode laser at 300 m W through thinning. The laser thinning will be performed by making 2-3 holes without reaching the inner membrane at a depth of60-80% of the Zona pellucida thickness.
  Arms: Zona pellucida thinning
Procedure: Zona pellucida drilling — Laser-assisted hatching will be conducted using a Laser System with a 1.48-μm diode laser at 300 m W through drilling. The laser opening will be made from the outside to the inside of the Zona pellucida.
  Arms: Zona pellucida drilling

SUMMARY:
Two hundred cycles will be enrolled (100 laser-assisted thinning and 100 laser-assisted drillings).

They will be compared regarding the implantation and clinical pregnancy rates

DETAILED DESCRIPTION:
Two hundred cycles will be enrolled (100 laser-assisted thinning and 100 laser-assisted drillings).

All study participants will undergo controlled ovarian stimulation by GnRH agonist long protocol starting from mid-luteal phase. The complete pituitary suppression will be confirmed by serumE2 level less than 30 pg/ml and serum LH level less than 2 mIU/ml, then gonadotropin therapy will be started from day 2 to the day of maturation confirmed by the presence of 3 mature follicles or more, one of them 18 mm; at this time 10000 IU of hCG will be administered then ovum pick up done 36 hours after hCG administration under transvaginal ultrasound guidance Cumulus cell masses around the oocytes will be removed using pull-and-cut denudation pipettes in a 5-well culture dish (MTG, Bruckberg, Germany) containing 27 IU/mL of hyaluronidase.

All oocytes that will be mature at 4-6 h after oocyte collection will be inseminated according to the quality of the spermatozoa and oocytes and the patient's previous IVF history. Fertilization will be confirmed 17-18 h after insemination by the presence of two distinct pronuclei. Zygotes will be cultured in 30-μL micro-drops with a 1-step medium and overlaid with paraffin oil in an atmosphere of 6% CO2, 5%O2, and 95% humidity at 37 °C. The available embryos will be assessed in all patients according to the criteria of equal and regular blastomeres, a viable blastomere number, and fragmentation ratio.

LAH will be conducted using a Laser System with a 1.48-μm diode-laser at 300 m W through thinning or drilling. The embryos will undergo either LAT or LAD in 10- to 20-μL micro-drops consisting of G-MOPS plus medium. The embryos will be fixed in the micro-drops on the inverted microscope. The size of one laser shot will be 5μm in the ZP using the same total number of 3000-μs pulses. In LAT, the goal of the thinning method is to make the outer portion of the outer protective glycoprotein layer thinner. The laser thinning will be performed by making 2-3 holes without reaching the inner membrane at a depth of60-80% of the ZP thickness. In LAD, the laser opening will be made from the outside to the inside of the ZP.

The laser beam shot towards the ZP above the perivitelline space between two blastomeres to minimize the risk of harming the embryo, under careful control. The embryos in the micro-drop will be washed several times after LAH and then transferred to a 1-well dish (Falcon 353,653, USA) containing G-2 culture medium. LAH was performed 2 to 3 h before embryo transfer. The embryos will be cultured in an atmosphere of 6% CO2, 5% O2, and 95% humidity at 37 °C.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a previous ICSI failure, unexplained infertility or male infertility

Exclusion Criteria:

* Patients with hydrosalpinx, pyosalpinx, endometriosis, or uterine fibroids

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | at 6 weeks of pregnancy
  Implantation rate = the total number of early gestational sacs/the total number of transferred embryos × 100%.

SECONDARY OUTCOMES:
Clinical pregnancy rate | at 6 weeks of pregnancy
  Clinical pregnancy rate = the number of pregnancy cycles/the total number of transfer cycles × 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ayoub, Principal Investigator — National Research Centre, Egypt
Locations (1):
- Private IVF Center, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No